CLINICAL TRIAL: NCT06433804
Title: Exploring the Clinicopathological Parameters of HER2 Low Breast Cancers
Brief Title: Clinicopathological Parameters of HER2 Low Breast Cancers
Status: Completed | Type: Observational
Sponsor: Vardhman Mahavir Medical College And Safdarjung Hospital (Other)
Responsible Party: Principal Investigator, SANA AHUJA, ASSISTANT PROFESSOR, Vardhman Mahavir Medical College And Safdarjung Hospital
Other Study IDs: CC-229
Record Dates: First submitted 2024-05-16; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: HER2 Low Breast Cancers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HER2 low
  Interventions: Diagnostic Test: HER2 IHC
- HER2 negative
  Interventions: Diagnostic Test: HER2 IHC

INTERVENTIONS:
Diagnostic Test: HER2 IHC — Immunohistochemistry for HER2

SUMMARY:
This was a retrospective cohort study which included all histologically proven cases of breast cancer in the 2 years from January 2022- December 2023 at a tertiary care centre.

This study was performed in line with STROCSS criteria. The following clinicopathological data was retrieved from the histopathological records- age, tumor size, nodal involvement, lymphovascular/ perineural invasion, and Bloom Richardson grading.

Routine histopathological processing was done followed by immunohistochemical analysis for ER, PR, HER2, Ki67 and AR. All the cases were categorised into Luminal A, B, Her2 enriched and triple-negative breast cancer based on the surrogate molecular classification. Further, all the cases were categorised into HER2 negative (no staining or incomplete weak membrane staining in ≤10% tumor cells), HER2 3+ (complete membranous staining) and HER2 low (1-2+ staining without amplification on ISH) based on consensus of two pathology consultants. The present study aims to evaluate the clinicopathological parameters of the HER2 low breast cancers.

ELIGIBILITY:
Inclusion Criteria:

* All histologically proven cases of breast cancer in the 2 years from January 2022- December 2023

Exclusion Criteria:

* Benign breast tumors

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All histologically proven cases of breast cancer in the 2 years from January 2022- December 2023
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Age (in years) | JANUARY 2022- DECEMBER 2023
  It will be measured for HER2 low breast cancer patients
Tumor stage (categorised from T1-T4) | JANUARY 2022- DECEMBER 2023
  This denotes status of stage of tumor- T1, T2, T3, T4. It will be measured for HER2 low breast cancer patients
N stage (categorised from N0-N3) | JANUARY 2022- DECEMBER 2023
  This denotes status of nodal involevement- N0, N1, N2 or N3. It will be measured for HER2 low breast cancer patients
Tumor grade (categorised from G1-G3) | JANUARY 2022- DECEMBER 2023
  This denotes whether tumor is well, modeartely or porrly differentiated. It will be measured for HER2 low breast cancer patients.
Surrogate molecular classification (Categorised as luminal/ triple negative) | JANUARY 2022- DECEMBER 2023
  This denoted the molecular classification of breast cancer based on ER, PR, Her2 expression.
Androgen receptor expression (Denoted as present or absent) | JANUARY 2022- DECEMBER 2023
  This denoted the immunohistochemical expression of androgen receptor which would be evaluted in all cases of HER2 low breast cancer

CONTACTS AND LOCATIONS:
Locations (1):
- VMMC SJH, New Delhi, India

IPD SHARING:
Plan to Share IPD: No